CLINICAL TRIAL: NCT04949945
Title: Efficacy of CBT on Positive Health Outcomes of Chronic Heart Failure Patients With Depression: A Randomized Controlled Trial
Brief Title: Efficacy of CBT on Positive Health Outcomes of Chronic Heart Failure Patients With Depression
Acronym: CaCBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Islamia University of Bahawalpur (Other)
Responsible Party: Principal Investigator, Saima Dastgeer, Student of PhD of Applied psychology, Islamia University of Bahawalpur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IslamiaB
Record Dates: First submitted 2021-06-03; First posted 2021-07-02 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Chronic Heart Failure; Depression
Keywords: Chronic Heart Failure; Depression; Self Help Culturally Cognitive Behavioral Therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHF patients who will receive guided self help culturally adapted cognitive behavioral therapy (Experimental): CHF(Chronic heart failure patients)(experimental group) will receive guided self help culturally adapted cognitive behavioral therapy.
  Interventions: Behavioral: Self Help Culturally Cognitive Behavioral Therapy
- CHF patients will not receive guided self help culturally adapted cognitive behavioral therapy (No Intervention): CHF(Chronic heart failure patients) (control group) will not receive Self Help Culturally Cognitive Behavior Therapy.

INTERVENTIONS:
Behavioral: Self Help Culturally Cognitive Behavioral Therapy — Experimental group (CHF patients)will be screened on PHQ9 questionnaire for depression after receiving guided self help culturally adapted cognitive therapy they will be reassessed for their depression,improvement in functional disability ,improvement in classification of NYHA,reduction in hospital admission as compare to control group.
  Arms: CHF patients who will receive guided self help culturally adapted cognitive behavioral therapy

SUMMARY:
The purpose of the study is to know the efficacy of Cognitive Behaviour Therapy on Positive Health Outcomes of Chronic Heart Failure Patients with Depression. It is a Randomized Control Trial (RCT) in which patients will be selected through purposive sampling techniques. Ages of patients will be 18-60 years. Data will be collected at outpatient department (OPD) of Ch.Pervaiz Elahi Institute of Cardiology Multan.Total measured sample size is 70 calculated by using G*Power 3.1.9.4.Patients will be randomized into Interventional and Control group, with 1:1 allocation, 35 patients in each group by virtual randomization(www.randomization.com). Diagnosed patients of heart failure for 6 or more than 6 months duration, EF ≤ 40 % on Trans Thoracic Echocardiography, patients with NYHA Heart Failure class II and III, patients with "mild" to "severe" level of depression based on PHQ-9 .Patients with other Psychiatric Disorders except depression, any substance dependence, mentally retarded, having personality disorders, already have received any psychotherapy or any psychiatric medication will be excluded. Patients will be assessed for functional disability by WHODAS 2.0 and severity of Heart Failure will be assessed by a Cardiologist using NYHA Heart Failure classification. Patients in experimental group will receive treatment as usual (TAU) and culturally adapted Cognitive Behavior Therapy. Patients in control group will receive treatment as usual (TAU) by a Cardiologist .

The aim of this experimental study is to study the efficacy of culturally adapted Cognitive Behavioral Therapy in patients with chronic heart failure with depression. To study the above-mentioned phenomenon, following hypotheses are formulated:

Hypothesis 1:

Patients receiving culturally adapted Cognitive-Behavioral Therapy will show reduction in their level of depression than patients not receiving intervention.

Hypothesis 2:

Patients will improve in NHYA heart failure class, by receiving CaCBT in experimental group as compared to control group.

Hypothesis 3:

Patients who will receive CaCBT will show less repeated Hospitalization in experimental group as compared to control group.

Hypothesis 4:

Patients in the intervention group will show betterment in the functional disability from pretest to post-test as compared to non- interventional group.

ELIGIBILITY:
Inclusion Criteria:

Chronic heart failure patient will be assessed by the following inclusion criteria; patients with

1. Diagnosed heart failure patients for 6 and more than 6 months duration,
2. EF < 40 % on Echocardiography ,
3. class II and III of NYHA heart failure,
4. "mild" to "severe" depression based on patients health questionnaire 9
5. who can understand, read, and write in Urdu will be included in study.

Exclusion Criteria:

Chronic heart failure patient will be assessed by the following exclusion criteria; patient with

1. any psychiatric disorders except depression,
2. substance dependence, mental retardation, personality disorders,
3. who have had received any psychotherapy or any psychiatric medication,
4. who are not willing to continue the sessions anymore, and the absence in more than two sessions will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-10 (Estimated); Study Completion 2021-11-29 (Estimated)

PRIMARY OUTCOMES:
change in scores of depression measured by patients' health questionnaire 9 | change from baseline scores of depression at 2 and half months of intervention in experimental and control group.
  change in scores of depression will be measured by Patients' Health Questionnaire 9. The PHQ-9 total score ranges from 0 to 27 (scores of 0- 4 are classified as none,5-9 mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; 20-27 as severe depression )from baseline to 2 and half months of intervention in control and experimental group.

SECONDARY OUTCOMES:
change in functional disability by world health organization disability assessment schedule II version. | Change in functional disability scores by world health organization disability assessment schedule II version will be measured from baseline to 2 and half months of intervention in control and experimental group.
  change in functional disability scores in control and experimental group by world health organization disability assessment schedule II version from baseline to 2 and half months of intervention in control and experimental group. It has 12 items for each item the patient has five choices; the score, depending on the choice, ranges from 0 (none) through to 4 (extreme). Therefore, the total score ranges from 0 to 48 points, with higher scores indicating higher functional disability. The score is expressed in percentage (divided by 48 and multiplied by 100 ) .The severity of functional disability is based on the calculated percentage as follows: none (0-4%), mild (5-24%), moderate (25-49%), severe (50-95%), and complete (96-100%) .
Change in New York Heart Association Classification of patients by a consultant cardiologist. | Change in class of New York Heart Association Classification of patients at 2 and half months of intervention and will be measured by a consultant cardiologist on New York Heart Association Classification in experimental and control group.
  Change in class of patients measured by a consultant cardiologist on New York Heart Association Classification( The New York Heart Association functional class was categorized into four classification system of physical functioning which is ranged from I no symptoms that have an impact on ordinary daily activities to IV symptoms occur at rest
  )in experimental and control group after 2 and half months of intervention .
Change in number of repeated hospitalization by patients' feedback. | Change in experimental group's number of repeated hospitalization compared to control group's repeated number of hospitalization after 2 and half months of intervention.
  Change in number of repeated hospitalization of experimental group will be measured by patients' feedback comparing with control group's repeated numbers of hospitalization after 2 and half month of intervention .

CONTACTS AND LOCATIONS:
Locations (1):
- Chauhdary Pervaiz Ellahi Institute of Cardiology, Multan, Punjab Province, Pakistan